CLINICAL TRIAL: NCT01477060
Title: Modulation of Response to Hormonal Therapy With Lapatinib and/or Metformin in Patients With HER2-negative, ER and/or PgR Positive Metastatic Brest Cancer With Progressive Disease After First-line Therapy
Brief Title: Modulation of Response to Hormonal Therapy With Lapatinib and/or Metformin in Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to insufficient accrual
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROLT/02; 2011-000155-16 (EudraCT Number)
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM A - Lapatinib (Other): hormonal therapy + lapatinib (1250mg/die) until disease progression or extraordinary medical circumstances occur or intolerable toxicities occur or the patient withdraws consent.
  Interventions: Drug: Lapatinib
- ARM B - Metformin (Other): Hormonal therapy + metformin until disease progression or extraordinary medical circumstances occur or intolerable toxicities occur or the patient withdraws consent.
  Interventions: Drug: Metformin
- ARM C - Lapatinib + Metformin (Other): Hormonal therapy + lapatinib + metformin until disease progression or extraordinary medical circumstances occur or intolerable toxicities occur or the patient withdraws consent.
  Interventions: Drug: Lapatinib; Drug: Metformin

INTERVENTIONS:
Drug: Lapatinib — 1250 mg/ die, os
  Arms: ARM A - Lapatinib; ARM C - Lapatinib + Metformin
Drug: Metformin — 1500 mg/die, os
  Arms: ARM B - Metformin; ARM C - Lapatinib + Metformin

SUMMARY:
Target Population: female patients with HER2-negative, ER and/or PgR positive breast cancer in progression after first-line hormonal therapy.

The study rationale is based on the potentiality of reversing endocrine-resistance by Lapatinib

* Activity on compensatory-adaptive mechanisms of hyperactivity of signals generated by HER2 family
* Modulation of energy balance and signals associated to survival through AMPK activation (via Calmodulin) Metformin
* Indirect mechanism, through reduced insulin receptors and IGFR stimulation, with reduces proliferative effects downstream
* Direct mechanism, through AMPK activation (via LKB1), with reduced protein synthesis (mTOR inhibition) and increased availability of intracellular energy Lapatinib and Metformin
* AMPK "Double"activation, through different potentially additional mechanisms.
* Inhibition of proliferative mechanisms for interference on various intracellular target

  * IR (A e/o B); IGFR
  * EGFR; HER2

Primary objectives :

1. To assess the rate of patients free from disease progression at 3 months from randomization

Secondary objectives :

1. To assess the overall response rate
2. To assess the duration of response
3. To assess 3-years overall survival rate
4. To assess tolerability of each proposed treatment Female patients with HER2-negative, ER and/or PgR positive breast cancer in progression after first-line hormonal therapy will randomized to receive: hormonal therapy + lapatinib or hormonal therapy + metformin or hormonal therapy + metformin + lapatinib with a ratio 1:1:1.

For each arm of the study the following sample size is required:

* First step: 23 patients, for a total of 69 patients in all 3 arms
* Second step: further 33 patients, for a total of 168 patients in all 3 arms.

DETAILED DESCRIPTION:
Treatment Plan Patient will continue to be treated with the same hormone therapy at the same dose, route and schedule

Patients will be randomized to receive:

A: Lapatinib, 1250 mg/die, os B: Metformin, 1500 mg/die, os C: Lapatinib + Metformin, 1250 mg+1500 mg/die, os Patients will receive study treatment until disease progression is documented, extraordinary medical circumstances occur, intolerable toxicities occur, or the patient withdraws consent

Statistical consideration Randomization will be stratified according to the site of metastases: visceral versus non-visceral lesions. The primary objective of this study is to evaluate the rate of patients free of disease progression at 3 months from randomization. The final analysis of this objective will be conducted when a total of 168 patients are enrolled across the three arms. This is the number of patients needed for a test with an experiment-wise alpha = 0.05 and power = 80% to show a statistically significant increment of 10% to the rate of patients without disease progression at 3 months, assuming a rate of 5% for treatments without lapatinib and/or metformin (P0=5% and P1=15%). After having accrued a total of 23 evaluable patients in each arm, the trial design can proceed to step 2 randomizing additional patients to each arm only if two or more patients are free of disease progression at 3 months. Otherwise, the study arm with less than expected responses will be discontinued. In the second stage 33 additional patients will be enrolled in each study arm to reach a total of 56 total patients per arm. If less than 6 patients per arm will be free of disease progression then the increment of corresponding treatment will be considered not significant.

Procedures:

The study will consist of a screening period, a treatment period and follow up for survival Screening Phase

Within 4 weeks prior randomization:

A signed written, informed consent will be obtained prior to any study specific assessments are initiated. The following will be performed prior to randomization

* Radiographic complete assessment of disease status (chest Xray; liver ultrasound, bone scan and CT or MR of target lesions and involved sites)
* Hematology and biochemistry
* Pregnancy test for women of child-bearing potential
* Cardiac assessment with ECG, echocardiography or multi-gated scintigraphic scan (MUGA)
* Medical history, physical examination, vital signs, signs and symptoms of breast cancer lesions, weight, height, ECOG performance status

Treatment Phase:

MONTHLY up to 3 months since randomization

* Physical examination, including clinical disease assessment, ECOG performance status, vital signs
* Hematology and biochemistry
* Safety evaluation (i.e. routine collection of adverse events)
* Patient's compliance
* Concomitant therapy

EVERY 3 MONTHS after the first 3 months of treatment until disease progression is documented, intolerable toxicities occur, or the patient withdraws consent:

* Physical examination, including clinical disease assessment, ECOG performance status, vital signs
* Radiographic disease assessment (using the same methods at screening)
* Hematology and biochemistry
* Safety evaluation (i.e. routine collection of adverse events)
* Concomitant therapy
* Patient's compliance

EVERY 6 MONTHS until disease progression is documented, intolerable toxicities occur, or the patient withdraws consent:

* Complete radiographic assessment
* Assessment of the LVEF using the same method at screening

Afterwards:

EVERY 6 MONTHS after disease progression or trial discontinuation due to intolerable toxicities or other reasons. Patients may receive other therapy following study discontinuation. Patients will continue to be followed for survival for a minimum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a histologically or cytologically confirmed adenocarcinoma of the breast progressing from prior hormonal therapy
2. Receptor positive disease (ER+ and/or PgR+)
3. HER2 negative
4. Pre- and post-menopausal status
5. Documented disease progression after first-line hormone therapy
6. Age ≥18 years.
7. Measurable or evaluable metastatic disease
8. Life expectancy > 3 months
9. ECOG Performance Status < 1
10. Adequate bone marrow, liver, and renal function as assessed by the following parameters:

    * Hemoglobin > 9.0 g/dl
    * Leucocytes count ≥ 3,000/mL
    * Absolute neutrophil count (ANC) ≥ 1.500/mL
    * Platelet count ≥ 100,000/mL
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement)
    * Albumine and total bilirubin ≤ 1.5 x ULN
    * Prothrombin Time (PT) < 70 %
    * Serum creatinine < 1.4 mg/ml, creatinine clearance > 70 ml/min
11. Normal Respiratory Function and Saturation level ≥ 90%
12. New York Hearth Association (NYHA) Classification ≤ 2 and baseline left ventricular ejection fraction (LVEF)≥ 50%
13. Patients must be willing and able to sign a written informed consent.

Exclusion Criteria:

1. Previous or concomitant treatment with lapatinib and/or metformin
2. More than one line of prior hormone therapy for metastatic breast cancer.
3. More than two lines of prior chemotherapy for metastatic breast cancer
4. Unique location of disease local-regionally treated (surgery, radiotherapy , other)
5. Disease progression not documented or less than 30%
6. Metastatic disease defined as aggressive at investigator's judgement (e.g. visceral disease more than >1/3 of involved parenchyma, symptomatic disease requiring intensive supportive measures or therapies not allowed by protocol)
7. Patients with brain metastasis
8. Osteosclerotic bone metastasis as unique disease site
9. Pathological tumor markers as unique sign of progressive disease
10. Concomitant treatment with any other anticancer drugs (biphosphonates are permitted)
11. Serious, not solved or unstable toxicity from previous treatment
12. Diabetes mellitus Type I and Type II
13. Renal insufficiency (creatinine ≥ 1.4 mg/ml)
14. Malabsorption syndrome or diseases that significantly may alter gastroenteric functions
15. Other serious illness or medical conditions judged by the investigator to be clinically significant that may adversely affect patient's participation in the trial or interfere with safety profile
16. Active clinically significant or uncontrolled infections (bacterial or viral)
17. Known history of unstable angina (angina symptoms at rest), cardiac ventricular arrhythmias clinically significant, myocardial infarction, stroke or congestive heart failure within 12 months prior to randomization
18. History of lactic acidosis
19. Evidence or symptoms of hepatic insufficiency
20. Chronic alcoholism
21. Concomitant treatment with amiodarone or any other agent that could interfere with study drugs
22. Known or suspected hypersensitivity or allergy to lapatinib, metformin or used excipients
23. Women who are pregnant or lactating
24. History of previous cancer, unless at low risk of relapse per investigator's judgement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of patients free from disease progression | 3 months from randomization

SECONDARY OUTCOMES:
overall response rate | 3 years
Progression Free Survival | 3 years
Time to progression | 3 years
Overall survival | 3 years
  To assess 3-years overall survival rate
Number of participants with toxicities as a measure of tolerability of each proposed treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Milvia Zambetti, MD, Principal Investigator — Ospedale San Raffaele
Locations (11):
- Italy (11):
  - Cliniche Gavazzeni S.p.A. - Humanitas Gavazzeni, Bergamo, BG
  - Fondazione Poliambulanza, Brescia, BS
  - Azienda Ospedaliera San Gerardo, Monza, MB
  - Azienda Ospedaliera "G. Salvini" - P.O. Garbagnate Milanese, Garbagnate Milanese, MI
  - Ospedale Civile Di Legnano, Legnano, MI
  - IRCCS Fondazione San Raffaele Monte Tabor, Milan, MI
  - IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Azienda Ospedaliera Ospedale Ca' Granda, Milan, MI
  - Fondazione Salvatore Maugeri Clinica del Lavoro e della Riabilitazione - Reparto Riabilitazione Oncologica, Pavia, PV
  - Fondazione Salvatore Maugeri Clinica del Lavoro e della Riabilitazione - U.O. Oncologia, Pavia, PV
  - Azienda Ospedaliera della Valtellina e della Valchiavenna - P.O. Sondrio, Sondrio, SO